CLINICAL TRIAL: NCT00188955
Title: Phase 4 Randomized, Controlled Study Comparing Sirolimus and Mycophenolate Mofetil to Prevent or Reverse Progression in Pediatric Renal Transplants With Chronic Allograft Nephropathy
Brief Title: Pilot Study on the Use of Sirolimus to Treat Chronic Allograft Nephropathy in Children After Kidney Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WINNIPEG-CAN-1
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Kidney Transplantation
Keywords: pediatric; chronic allograft nephropathy; chronic rejection; interstitial fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Sirolimus

INTERVENTIONS:
Drug: sirolimus

SUMMARY:
The purpose of this study is to determine whether treatment with sirolimus, in combination with low-dose tacrolimus and prednisone, is effective for the treatment of chronic allograft nephropathy (progressive scarring) in children who have previously received a kidney transplant. This treatment is compared to the standard therapy which uses low-dose tacrolimus, mycophenolate mofetil and prednisons.

This study is a pilot study that will determine whether treatment with sirolimus reduces or improves the rate of scarring seen on kidney biopsy of the transplanted kidney over time, compared to children who continue to be treated with mycophenolate mofetil.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Title Of Study: A Single Center, Prospective, Randomized, Controlled Study Of Two Chronic Immunosuppressive Protocols Using Sirolimus Or Mycophenolate Mofetil To Prevent Or Reverse Disease Progression In Pediatric Renal Transplants With Chronic Allograft Nephropathy

Short Title: Winnipeg-CAN-1

Clinical Trial: Phase-IV

Objectives: This prospective, randomized, controlled study will evaluate the effectiveness of two different chronic immunosuppressive protocols in the treatment of chronic allograft nephropathy (CAN) in children. One protocol will continue with standard immunosuppression which includes mycophenolate mofetil (MMF), and the other will substitute MMF with sirolimus.

The primary objective is as follows:

· To evaluate the effectiveness of treatment with sirolimus in pediatric renal transplant recipients with established CAN compared to MMF at reducing the rate of progression of CAN as measured by prospective histological evaluation of sequential kidney biopsies using quantification of interstitial fibrosis by image analysis and a validated standardized scoring schema (Banff 97 criteria).

The secondary objectives are as follows:

* To evaluate the effectiveness of treatment with sirolimus in pediatric renal transplant recipients with established CAN compared to MMF at slowing the rate of clinical deterioration associated with progression of CAN as measured by the change of serum creatinine and corrected glomerular filtration rate (GFR) over the study period.
* To analyze the effect of treatment with sirolimus in pediatric renal transplant recipients with established CAN compared to MMF on the incidence of late AR as identified by prospective histological evaluation of sequential kidney biopsies.
* To analyze the effect of treatment with sirolimus in pediatric renal transplant recipients with established CAN compared to MMF on the incidence graft failure as defined by a return to dialysis, re-transplantation or death from uremic complications.
* To analyze the differences in the expression of molecular markers of fibrosis in pediatric renal transplant recipients with established CAN treated with sirolimus compared to MMF by immunohistochemical identification of extracellular matrix protein expression and remodeling and quantification by image analysis.

Study Design: The study will be a prospective, single-centre, randomized, controlled trial in pediatric patients with functioning kidney transplants who have biopsy-proven CAN. The study is designed to compare the efficacy of two chronic immunosuppression regimens intended for the treatment of CAN. Patients (aged 1-17 years) who have CAN demonstrated on protocol biopsy or on biopsy done for clinical suspicion of CAN, will be considered for enrollment. Eligible patients will be enrolled and treatment will be randomized between one of two treatment groups: Group A will receive sirolimus in combination with low-dose tacrolimus and prednisone; Group B will receive the current local standard therapy, which is MMF, low-dose tacrolimus and prednisone. All other transplant care will be according to standard local practice.

Study participants will be followed for a period of 2 years, and will undergo protocol biopsies at 1 and 2 years. The timing of these biopsies will coincide with already planned protocol biopsies. Clinical, laboratory and histological data will be gathered prospectively to determine efficacy according to pre-defined criteria measuring the extent of CAN and interstitial fibrosis. Study visits will coincide with routine clinic visits, except for weekly visits at the study onset to titrate drug dosing according to trough levels. Blood and urine tests, blood pressure monitoring, timed urine collections and nuclear GFR testing will be performed according to the normal clinical care protocols. Additional pharmacokinetic testing will occur at 3 and 12 months.

Participants will be enrolled over a 2-year period and will be followed according to study protocol for 2 years. 40 patients will be enrolled.

Dosages, Route and Dose Regimen:

Patients randomized to Group A will receive an initial oral loading dose of sirolimus 3 mg/m2 in 2 divided doses (1.5 mg/m2/dose bid) on study day 1. Beginning on study day 2, patients will receive 1mg/m2/day orally in divided doses (0.5 mg/m2/dose) every 12 hours. Therapeutic drug monitoring of 12-hour trough concentrations will be performed at weeks 1-4, then monthly for the first 3 months, then at least every 3 months, and dose adjustments will be made in order to achieve 12-hour trough levels between 8 ng/ml and 12 ng/ml.

Patients randomized to Group B will continue to receive MMF 1200 mg/m2/day orally in divided doses (600 mg/m2/dose) every 12 hours starting on Study Day 1. Therapeutic drug monitoring of 12-hour trough concentrations will be performed at weeks 1-4, then monthly for the first 3 months, then at least every 3 months, and dose adjustments will be made in order to achieve 12-hour trough mycophenolic acid (MPA) levels of between 2.0 mg/ml and 4.0 mg/ml.

Safety Measurements:

Safety will be determined by monitoring AEs, vital signs, and laboratory parameters (clinical chemistry, hematology, and urinalysis) during the follow-up period. In particular, signs and symptoms associated with known medication side effects such as infection, malignancy, anemia (sirolimus), thrombocytopenia (sirolimus), hyperlipidemia (sirolimus), leukopenia (MMF) and GI effects (MMF). Serial monitoring of renal function will indicate acute rejection or drug toxicity, to be confirmed on biopsy.

Primary Efficacy And Secondary Endpoints:

Quantitative changes in CAN will be used to determine efficacy. Protocol renal allograft biopsies will be performed at 12 and 24 months after study enrollment and will be compared to the baseline histology obtained from routine protocol surveillance biopsy during the screening period which are performed at 1, 3, 6 12 months post-transplant, and yearly thereafter. The amount of CAN will be measured by semi-quantitative scoring of histological changes characteristic of CAN according to the Banff 97 schema, and interstitial fibrosis will be quantified using image analysis.

Secondary endpoints include changes of renal function, proteinuria, rates of acute rejection, graft survival, and the expression of proteins important in interstitial matrix remodelling by immunohistochemistry. Renal function will be monitored at each clinical visit and will be compared with baseline function over the duration of the study. In addition, quantitative assessment of GFR corrected for body surface area will be obtained at baseline, 1 and 2 years, by nuclear GFR measurement. Proteinuria will be quantified by 24-hour urine collection at baseline and every 6 months during the study or by spot protein:creatinine ratio.

Statistical Analysis:

Data are expressed as mean ± standard deviation. Quantitative TFR will be compared between groups using the change in TFR over time (DTFR) and the percent change from baseline (%DTFR). The Student's t-test will be used to compare the change between groups for the primary endpoint. One-way ANOVA will be used to detect significant change for multiple time-points, and multiple ANOVA to examine correlation between interval variables. Multiple regression analysis is used to determine the predictive value of different, possibly independent quantitative variables. Non-parametric variables will be analyzed using the Wilcoxon Signed Rank Test, and treatment differences over time using the Quade test. A difference of <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All male or female patients aged less than 17 years.
* The patient has undergone a kidney transplant, from a cadaveric or living donor with compatible ABO blood type.
* The patient is more than 12 months post-transplantation.
* The allograft demonstrates histological changes consistent with CAN according to the Banff 97 classification schema (minimum of ct1 and ci1 score for tubular atrophy and interstitial fibrosis respectively).

Exclusion Criteria:

* The patient, or in case the patient is minor, the patient's parent(s) or their legal representative, has been fully informed and will not give informed consent to participate in the study.
* The allograft demonstrates histological changes at the time of enrollment consistent with acute allograft rejection Grade Ia or worse, according to the Banff 97 classification schema (minimum of t2 and i2 score for tubulitis and interstitial inflammation respectively).
* The patient is known to be allergic or intolerant to MMF, sirolimus or any of their known metabolites.
* The patient for who routine protocol kidney biopsy is contraindicated.
* Patients whose maintenance immunosuppression does not include both tacrolimus and prednisone at the time on study enrollment.
* Patients previously treated with sirolimus.
* The patient requires ongoing dosing with a systemic immunosuppressive drug at study entry for any reason other than kidney transplantation.
* The patient and/or donor is known to be HIV or HCV positive.
* The patient has significant liver disease, defined as having during the past 28 days continuously elevated ASAT (SGOT) and/or ALAT (SGPT) levels greater than 3 times the upper value of the normal range of the investigational site.
* The patient has persistent leukopenia (WBC <3.0 x109/L).
* The patient has persistent thrombocytopenia (<100 x109/L).
* The patient has pre-existing significant hyperlipidemia (total cholesterol >7.8 mmol/L), not responding to medical therapy.
* The patient has pre-existing elevated triglycerides, not responding to medical therapy.
* The patient with malignancy or history of malignancy except for successfully treated Wilm's tumor (2 years) or non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* The patient has significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting or active peptic ulcer.
* The patient has previously received or is receiving an organ transplant other than kidney.
* The patient is taking or has been taking an investigational drug in the past 28 days or is currently participating in another clinical intervention trial.
* Patients with the relapsing, non-diarrheal form of haemolytic-uraemic syndrome.
* The patient is unlikely to comply with the protocol.
* The patient has any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may invalidate communication with the investigator
* Sexually active female patients who are pregnant or lactating or who do not consent to effective birth control.
* The patient is less than 6 years of age.
* The patient has significant and persistent EBV activity as measured by PCR amplification from blood samples.
* The patient has a prior history of post-transplant lymphoproliferative disease.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-03; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
histological quantification of interstitial fibrosis at 2 years

SECONDARY OUTCOMES:
Renal function at 1 and 2 years.
Proteinuria at 2 years.
Freedom from acute rejection and graft loss over the 2 year study period.
Cumulative incidence and prevalence of adverse events and serious adverse events over the 2-year study period.

CONTACTS AND LOCATIONS:
Overall Officials: Tom D. Blydt-Hansen, MD, Principal Investigator — University of Manitoba, Manitoba Institute of Child Health
Locations (1):
- Children's Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Manitoba Institute of Child Health — http://www.mich.ca/
- See also: Children's Hospital in Winnipeg — http://www.goodbear.mb.ca/
- See also: University of Manitoba — http://www.umanitoba.ca